CLINICAL TRIAL: NCT00705549
Title: Feasibility and Efficacy of Molecular Analysis-Directed Individualized Therapy Based of Tumoral mRNA Levels of ERCC1, RRM1 and BRCA1 in Advanced Non-Small-Cell Lung Cancer
Brief Title: Individualized Therapy Based of Tumoral mRNA Levels of ERCC1, RRM1 and BRCA1 in Advanced Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.23
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Advanced; NSCLC; ERCC1; RRM1; BCRA1; Alimta; Gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Docetaxel; Vinorelbine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- 1 (Experimental): Gemzar/Cisplatin
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- 2 (Experimental): Taxotere/Cisplatin
  Interventions: Drug: Cisplatin; Drug: Docetaxel
- 3 (Experimental): Cisplatin/Navelbine metronomic
  Interventions: Drug: Cisplatin; Drug: Vinorelbine
- 4 (Experimental): Taxotere/Gemzar
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- 5 (Experimental): Gemzar
  Interventions: Drug: Gemcitabine
- 6 (Experimental): Taxotere
  Interventions: Drug: Docetaxel
- 7 (Experimental): Navelbine metronomic
  Interventions: Drug: Vinorelbine
- 8 (Experimental): Alimta/Cisplatin
  Interventions: Drug: Cisplatin; Drug: Pemetrexate
- 9 (Experimental): Alimta/Gemzar
  Interventions: Drug: Gemcitabine; Drug: Pemetrexate
- 10 (Experimental): Taxotere
  Interventions: Drug: Docetaxel
- 11 (Experimental): Alimta
  Interventions: Drug: Pemetrexate

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine I.V at the dose of 1000mg/m2 on Day 1 and Day 8
  Other Names: Gemzar
  Arms: 1; 4; 5; 9
Drug: Cisplatin — Cisplatin I.V at the dose of 75mg/m2 on Day 1
  Other Names: CDDP
  Arms: 1; 2; 8
Drug: Docetaxel — Docetaxel I.V at the dose of 75mg/m2 on Day 1
  Other Names: Taxotere
  Arms: 10; 2; 4; 6
Drug: Cisplatin — Cisplatin I.V at the dose of 80mg/m2 on Day 1
  Other Names: CDDP
  Arms: 3
Drug: Vinorelbine — Vinorelbine per os 50mg every Monday, Wednesday and Friday
  Other Names: Navelbine
  Arms: 3; 7
Drug: Pemetrexate — Pemetrexate I.V 500mg/m2 on Day 1
  Other Names: Alimta
  Arms: 11; 8; 9

SUMMARY:
This is a prospective pilot phase II trial, in patients with wet stage IIIb and IV NSCLC using chemotherapy regimens which will be defined according to the pharmacogenomic profile (tumoral expression of ERCC1, BRCA1 and RRM1) of the tumor cells.

DETAILED DESCRIPTION:
Advanced stage NSCLC is essentially a fatal disease and treatment is mainly palliative. Systemic cisplatin-based chemotherapy remains the mainstream for the treatment of advanced non-small cell lung cancer (NSCLC) since it improves survival, symptom control and quality of life compared to best supportive care.

The selection of appropriate treatment for individual patients remains a challenge in clinical oncology, particularly in the advanced disease. Several lines of evidence indicate that polymorphisms, gene transcripts and gene mutations can play a predictive role and can be used to tailor chemotherapy in different subgroups of cancer patients. There are evidence lead us to use the expression levels of ERCC1 by the tumor as a molecular marker for customized chemotherapy. Another gene, the BRCA1 has a crucial role in DNA repair, since it is implicated in transcription-coupled nucleotide excision repair (TC-NER), leading to radio- and chemo-resistance. RRM1,localized in 11p15.5,also acts as a putative tumor suppressor gene. RRM1 overexpression was related to gemcitabine resistance in human oropharyngeal epidermoid carcinoma KB cells as well as in patients with NSCLC. For those reason we decided to conduct a prospective pilot phase II trial, in patients with wet stage IIIb and IV NSCLC using chemotherapy regimens which will be defined according to the pharmacogenomic profile (tumoral expression of ERCC1, BRCA1 and RRM1) of the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven Stage IV and Stage III (with malignant pleural or pericardial effusion) squamous or adenocarcinoma carcinomas of the lung
* Adequate Formalin Fixed Paraffin Embedded tumor sample provided for molecular analysis
* No previous anticancer treatment for metastatic/advanced disease. Patients who received prior adjuvant chemotherapy are eligible if they have remained free of disease for at least 6 months after the completion of adjuvant therapy.
* Age above 18 years
* Performance status (ECOG) 0-2
* Life expectancy >= 3 months
* Effective contraception for both male and female subjects if the risk of conception exists
* Adequate hematologic parameters (absolute neutrophil count >= 1.5x109/L and platelets >= 100x109/L), creatinine (GFR>= 60ml/min) and total bilirubin < 1.5 times the upper limit of normal; aspartate and alanine aminotransferase < 2,5 times the upper limit of normal
* All patients will have to sign written informed consent in order to participate in the study

Exclusion Criteria:

* Patients with non-squamous tumors who have no contradiction for administration of bevacizumab
* Active infection or malnutrition (loss of more than 20% of the body weight)
* Known hypersensitivity reaction to any of the component of the treatment
* Concurrent or previous chronic systemic immune therapy
* Pregnancy (absence to be confirmed by ß-HCG test) or lactation period
* Known alcohol/drug abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent
* A second primary tumor other than non-melanoma skin cancer or in situ cervical carcinoma
* Previous radiotherapy to the target lesions. Patients treated with palliative radiotherapy had to have measurable metastatic disease outside the irradiation fields
* Patients with severe cardiac dysfunction, unstable angina petrosis, or high risk of uncontrolled arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) based on the pharmacogenomic profile of the ERCC1, RRM1 and BRCA1 expression | Objective responses confirmed by CT or MRI

SECONDARY OUTCOMES:
Determine the incidence of the different pharmacogenomic profiles as defined by the combined expression of ERCC1, RRM1 and BCRA1 | Comparison of molecular determinants for response in the primary tumor and peripheral blood (ERCC1 polymorphism ,TXR1 and TSP1 mRNA expression by Q-RT-PCR, Molecular markers related to responsiveness to Alimta )
Time to Tumor Progression | 1 year
Overall Survival | 1 year
Toxicity | Toxicity assessment on each chemotherapy cycles

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki